CLINICAL TRIAL: NCT02567253
Title: Intraoperative Intraperitoneal Chemoperfusion to Treat Peritoneal Minimal Residual Disease in Stage III Ovarian Cancer: A Randomized Phase II Trial
Brief Title: Intraoperative Intraperitoneal Chemoperfusion to Treat Peritoneal Minimal Residual Disease in Stage III Ovarian Cancer
Acronym: OvIP1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGO/2015/002
Record Dates: First submitted 2015-09-23; First posted 2015-10-02 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer
Keywords: Cytoreductive surgery; (H)ipec; Ovarian cancer; Cisplatin; Peritoneal carcinomatosis; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms | interventions — Cytoreduction Surgical Procedures; Cisplatin; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- low dose, normothermic (Experimental): CRS + normothermic (37°C) intraoperative intraperitoneal chemoperfusion, with 75mg/m² Cisplatin during 90min + adjuvant chemotherapy
  Interventions: Procedure: Cytoreductive surgery; Drug: IPEC with Cisplatin (75mg/m²)
- high dose, normothermic (Experimental): CRS + normothermic (37°C) intraoperative intraperitoneal chemoperfusion, with 100mg/m² Cisplatin during 90min + adjuvant chemotherapy
  Interventions: Procedure: Cytoreductive surgery; Drug: IPEC with Cisplatin (100mg/m²)
- low dose, hyperthermic (Experimental): CRS + hyperthermic (41°C) intraoperative intraperitoneal chemoperfusion, with 75mg/m² Cisplatin during 90min + adjuvant chemotherapy
  Interventions: Procedure: Cytoreductive surgery; Drug: Hypertherm IntraPEritoneal Chemotherapy with Cisplatin (75mg/m²)
- high dose, hyperthermic (Experimental): CRS + hyperthermic (41°C) intraoperative intraperitoneal chemoperfusion, with 100mg/m² Cisplatin during 90min + adjuvant chemotherapy
  Interventions: Procedure: Cytoreductive surgery; Drug: HIPEC with Cisplatin (100mg/m²)

INTERVENTIONS:
Procedure: Cytoreductive surgery — Complete or nearly complete (CC-0 or CC-1) macroscopic cytoreduction at the time of surgery of peritoneal carcinomatosis from ovarian cancer
Drug: IPEC with Cisplatin (75mg/m²) — Intraperitoneal normotherm (37°C) administration of Cisplatin (75mg/m²) , during 90min
  Arms: low dose, normothermic
Drug: IPEC with Cisplatin (100mg/m²) — Intraperitoneal normotherm (37°C) administration of Cisplatin (100mg/m²), during 90min
  Arms: high dose, normothermic
Drug: Hypertherm IntraPEritoneal Chemotherapy with Cisplatin (75mg/m²) — Intraperitoneal hypertherm (41°C) administration of Cisplatin (75mg/m²), during 90min
  Arms: low dose, hyperthermic
Drug: HIPEC with Cisplatin (100mg/m²) — Intraperitoneal hypertherm (41°C) administration of Cisplatin (100mg/m²), during 90min
  Arms: high dose, hyperthermic

SUMMARY:
The OvIP1 study is designed to examine how drug dose and perfusion temperature affect the pharmacokinetics and pharmacodynamics of cisplatin used as (hyperthermic) intraperitoneal chemoperfusion, as an adjunct to surgery, in women with stage III epithelial ovarian cancer.

DETAILED DESCRIPTION:
Stage III ovarian cancer (OC) remains an important cause of cancer related mortality in women. After successful initial treatment, most patients eventually develop recurrent peritoneal disease which can only arise from peritoneal minimal residual disease (pMRD) left after primary cytoreductive surgery (CRS). Intensification of locoregional therapy through intraoperative intraperitoneal chemoperfusion (IPEC) immediately following CRS may prevent or delay peritoneal recurrence. Although IPEC, usually under hyperthermic conditions, is increasingly used in OC, its efficacy and the potential benefit of hyperthermia are at present unknown.The primary aim of this study is to assess the pharmacokinetic and pharmacodynamic properties of IP cisplatin administered under normothermic or hyperthermic conditions, and at different dosing schedules. Additional endpoints include surgery related morbidity and mortality, quality of life, overall survival, disease free survival, peritoneal recurrence free survival, peritoneal cytology, and exploration of potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Tumor type:

  * Biopsy proven serous epithelial ovarian carcinoma or peritoneal carcinoma
* Primary or recurrent disease
* Extent of disease:

  * Positive retroperitoneal lymph nodes and /or microscopic metastasis beyond the pelvis (FIGO stage III, Appendix (47))
  * Stage IV with unilateral pleural fluid allowed
  * Complete or nearly complete macroscopic cytoreduction at the time of surgery (CC-0 or CC-1) deemed possible based on imaging, laparoscopy, or both
* Second-line patients; platinum sensitive
* Age over 18 years
* No major cardiac or respiratory disease
* Adequate performance status (Karnofsky index > 70%)
* Adequate mental faculty, allowing to understand the proposed treatment protocol and provide informed consent
* Expected life expectancy more than 6 months
* Laboratory data:

  * Serum creatinine ≤ 1.5 mg/dl or a calculated Glomerular Filtration Rate (GFR) (CKD-EPI) ≥ 60 mL/min/1.73 m2
  * Serum total bilirubin ≤ 1.5 mg/dl, except for known Gilbert's disease
  * Platelet count > 100.000/µl
  * Hemoglobin > 9g/dl
  * Neutrophil granulocytes > 1.500/ml
  * International Normalized Ratio (INR) ≤ 2
* Absence of alcohol and/or drug abuse
* No other concurrent malignant disease
* No inclusion in other clinical trials interfering with the study protocol
* No concurrent chronic systemic immune or hormone therapy, except neoadjuvant chemotherapy
* Absence of any severe organ insufficiency
* No pregnancy or breast feeding
* Written informed consent

Exclusion Criteria:

* Severe or uncontrolled cardiac insufficiency, including recent (< 6 months) occurrence of myocardial infarction, the presence of congestive cardiac insufficiency, of symptomatic angor in spite of optimal medical care, of cardiac arrhythmia requiring medical treatment presenting insufficient rhythm control, or uncontrolled arterial hypertension
* Pregnancy or breast feeding
* Platinum resistant or refractory disease
* Active bacterial, viral or fungal infection
* Active gastro-duodenal ulcer
* Parenchymal liver disease (any stage cirrhosis)
* Uncontrolled diabetes mellitus
* Severe obstructive or restrictive respiratory insufficiency
* Psychiatric pathology capable of affecting comprehension and judgment faculty
* Tumor in the presence of obstruction
* Evidence of extra-abdominal disease (with the exception of unilateral malignant pleural effusion) or extensive liver metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Tissue penetration distance of cisplatin in peritoneal tumor tissue nodules using laser-ablation inductively couples plasma mass spectrometry | 1 tumor nodule will be immediately fixed in liquid nitrogen after cytoreductive surgery and chemoperfusion. Frozen sections will be ablated through study completion
  This will be analyzed via laser ablation-inductively coupled plasma- mass spectrometry (LA-ICP-MS)

SECONDARY OUTCOMES:
Surgical morbidity and mortality will be measured using Dindo-Clavien classification | Within 30 days after surgery and intraoperative intraperitoneal chemoperfusion
  This will be estimated with the Dindo-Clavien classification
Cancer-specific Quality of Life-C30 | 3 weeks before operation, 6 weeks after and 3, 6, 12, 18 and 24 months after surgery and chemoperfusion
  This will be investigated using the cancer-specific (C30) European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaires
Disease-specific Quality of Life-OV28 | 3 weeks before operation, 6 weeks after and 3, 6, 12, 18 and 24 months after surgery and chemoperfusion
  This will be investigated using the disease-specific (OV28) European Organization for Research and Treatment of Cancer (EORTC) Quality of Life questionnaires
Maximum perfusate concentration (Cmax) of cisplatin | T=0min (before chemoperfusion), T=15min, T=30min, T=90min (during chemoperfusion); T=2h, T=3h, T=7.5h, T=24h (after start chemoperfusion)
  Cisplatin (free + bounded) will be measured in perfusate, using high performance liquid chromatography coupled to an inductively coupled plasma- mass spectrometry (HPLC-ICP-MS)
Maximum plasma concentration (Cmax) and Area Under The Curve (AUC) of cisplatin | T=0min (before chemoperfusion); T=15min, T=30min, T=90min (during chemoperfusion); T=2h, T=3h, T=7.5h, T=24h (after start chemoperfusion)
  Cisplatin (free + bounded) will be measured in plasma, using high performance liquid chromatography coupled to an inductively coupled plasma- mass spectrometry (HPLC-ICP-MS)
Pharmacodynamics (PD) of cisplatin will be analyzed by visualizing the amount of DNA double-strand breaks (dsb) via the specific DNA-adduct immunohistochemical Liedert staining | 1 tumor nodule will be immediately fixed in 4% paraformaldehyde and immunohistochemical stainings will be done through study completion
  PD of cisplatin will be studied via Pt-DNA adduct formation, using the Liedert staining which is specific for Pt-[Guanine, Guanine] adducts (Pt-[GG]) using Mab R-C18. The amount of double-strand breaks (dsb) will be analyzed then via fluorescence microscopy
Overall survival | 24 months after finishing the adjuvant chemotherapy
  Calculated from date of surgery until death
Disease free survival | 24 months after finishing the adjuvant chemotherapy
  Time interval between date of surgery and disease progression or death
Peritoneal recurrence free survival | 24 months after finishing the adjuvant chemotherapy
  Time interval between date of surgery and peritoneal recurrence or death
Expression analysis of selected biomarkers = Excision repair cross-complementation group 1 (ERCC1), Methylguanine methyltransferase enzyme (MGMT), Breast cancer gene 1 (BRCA1), Copper transporter 1 (CTR1) using quantitative PCR | 1 tumor nodule will be immediately fixed in liquid nitrogen. Histological coupes will be made through study completion
  Gene expression of potential predictive biomarkers using qPCR
Stromal composition and density of tumor tissues via analyzing collagen density, fibroblast Proliferation and DNA-intrastrand adduct formation of Pt-[GG] | 1 tumor nodule will be immediately fixed in 4% paraformaldehyde. Histological coupes will be made through study completion
  Analyzing collagen density using the sirius red staining, analyzing fibroblast proliferation using alfa smooth-muscle action (α-SMA) stainings and DNA intrastrand adduct formation of Pt-[GG] with the Liedert staining using Mab R-C18

CONTACTS AND LOCATIONS:
Overall Officials: Wim P Ceelen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- UZ Ghent, Ghent, East-Flanders, Belgium

REFERENCES:
- [Background] Coleman RL, Monk BJ, Sood AK, Herzog TJ. Latest research and treatment of advanced-stage epithelial ovarian cancer. Nat Rev Clin Oncol. 2013 Apr;10(4):211-24. doi: 10.1038/nrclinonc.2013.5. Epub 2013 Feb 5. PMID 23381004
- [Background] Foley OW, Rauh-Hain JA, del Carmen MG. Recurrent epithelial ovarian cancer: an update on treatment. Oncology (Williston Park). 2013 Apr;27(4):288-94, 298. PMID 23781692
- [Background] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Background] Markman M, Bundy BN, Alberts DS, Fowler JM, Clark-Pearson DL, Carson LF, Wadler S, Sickel J. Phase III trial of standard-dose intravenous cisplatin plus paclitaxel versus moderately high-dose carboplatin followed by intravenous paclitaxel and intraperitoneal cisplatin in small-volume stage III ovarian carcinoma: an intergroup study of the Gynecologic Oncology Group, Southwestern Oncology Group, and Eastern Cooperative Oncology Group. J Clin Oncol. 2001 Feb 15;19(4):1001-7. doi: 10.1200/JCO.2001.19.4.1001. PMID 11181662
- [Background] Alberts DS, Liu PY, Hannigan EV, O'Toole R, Williams SD, Young JA, Franklin EW, Clarke-Pearson DL, Malviya VK, DuBeshter B. Intraperitoneal cisplatin plus intravenous cyclophosphamide versus intravenous cisplatin plus intravenous cyclophosphamide for stage III ovarian cancer. N Engl J Med. 1996 Dec 26;335(26):1950-5. doi: 10.1056/NEJM199612263352603. PMID 8960474
- [Background] Jaaback K, Johnson N. Intraperitoneal chemotherapy for the initial management of primary epithelial ovarian cancer. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD005340. doi: 10.1002/14651858.CD005340.pub2. PMID 16437527
- [Background] Kyrgiou M, Salanti G, Pavlidis N, Paraskevaidis E, Ioannidis JP. Survival benefits with diverse chemotherapy regimens for ovarian cancer: meta-analysis of multiple treatments. J Natl Cancer Inst. 2006 Nov 15;98(22):1655-63. doi: 10.1093/jnci/djj443. PMID 17105988
- [Background] Ceelen WP, Van Nieuwenhove Y, Van Belle S, Denys H, Pattyn P. Cytoreduction and hyperthermic intraperitoneal chemoperfusion in women with heavily pretreated recurrent ovarian cancer. Ann Surg Oncol. 2012 Jul;19(7):2352-9. doi: 10.1245/s10434-009-0878-6. Epub 2009 Dec 29. PMID 20039210
- [Background] Issels RD. Hyperthermia adds to chemotherapy. Eur J Cancer. 2008 Nov;44(17):2546-54. doi: 10.1016/j.ejca.2008.07.038. Epub 2008 Sep 11. PMID 18789678
- [Background] Sun X, Li XF, Russell J, Xing L, Urano M, Li GC, Humm JL, Ling CC. Changes in tumor hypoxia induced by mild temperature hyperthermia as assessed by dual-tracer immunohistochemistry. Radiother Oncol. 2008 Aug;88(2):269-76. doi: 10.1016/j.radonc.2008.05.015. Epub 2008 Jun 5. PMID 18538874
- [Background] Bijelic L, Jonson A, Sugarbaker PH. Systematic review of cytoreductive surgery and heated intraoperative intraperitoneal chemotherapy for treatment of peritoneal carcinomatosis in primary and recurrent ovarian cancer. Ann Oncol. 2007 Dec;18(12):1943-50. doi: 10.1093/annonc/mdm137. Epub 2007 May 11. PMID 17496308
- [Background] Helm CW. The role of hyperthermic intraperitoneal chemotherapy (HIPEC) in ovarian cancer. Oncologist. 2009 Jul;14(7):683-94. doi: 10.1634/theoncologist.2008-0275. Epub 2009 Jul 16. PMID 19608639
- [Background] de Bree E, Helm CW. Hyperthermic intraperitoneal chemotherapy in ovarian cancer: rationale and clinical data. Expert Rev Anticancer Ther. 2012 Jul;12(7):895-911. doi: 10.1586/era.12.72. PMID 22845405
- [Background] Mulier S, Claes JP, Dierieck V, Amiel JO, Pahaut JP, Marcelis L, Bastin F, Vanderbeeken D, Finet C, Cran S, Velu T. Survival benefit of adding Hyperthermic IntraPEritoneal Chemotherapy (HIPEC) at the different time-points of treatment of ovarian cancer: review of evidence. Curr Pharm Des. 2012;18(25):3793-803. doi: 10.2174/138161212802002616. PMID 22591422